CLINICAL TRIAL: NCT02123368
Title: Treatment of Osteoarthritis by Intra-articular Injection of Bone Marrow Mesenchymal Stem Cells
Brief Title: Treatment of Knee Osteoarthritis by Intra-articular Injection of Bone Marrow Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMM/ART; 2009-017624-72 (EudraCT Number)
Record Dates: First submitted 2013-11-12; First posted 2014-04-25 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Mesenchimal stem cell; Knee
MeSH Terms: conditions — Osteoarthritis | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hialuronic acid (Active Comparator): Single intraarticular injection of Hyaluronic acid (Hyal One)
  Interventions: Drug: Hyaluronic acid
- Hyaluronic acid and MSC 10 (Active Comparator): Single intraarticular injection of Hyaluronic acid (Hyal One) 10 million Bone marrow mesenchimal stem cells
  Interventions: Drug: Hyaluronic acid; Biological: 10 million Bone marrow mesenchimal stem cells
- Hyaluronic acid AND MSC 100 (Active Comparator): Single intraarticular injection of Hyaluronic acid (Hyal One) 100 million Bone marrow mesenchimal stem cells
  Interventions: Drug: Hyaluronic acid; Biological: 100 million Bone marrow mesenchimal stem cells

INTERVENTIONS:
Drug: Hyaluronic acid — Single intraarticular injection of Hyaluronic acid (Hyal One)
  Other Names: HyalOne
Biological: 10 million Bone marrow mesenchimal stem cells — 10 million of Bone marrow mesenchimal stem cells
  Arms: Hyaluronic acid and MSC 10
Biological: 100 million Bone marrow mesenchimal stem cells — 100 million of Bone marrow mesenchimal stem cells
  Arms: Hyaluronic acid AND MSC 100

SUMMARY:
Purpose: To determine the safety, feasibility and effectiveness (clinical and radiological) of intra-articular administration of autologous mesenchymal stem cells (MSCs) in patients with knee osteoarthritis.

Patients and methods

Clinical trial phase I- II, randomized , multicenter , with three treatment arms and 10 patients for each group. The investigators compare the intraarticular injection of hialuronic acid against the administration of two different doses of mesenchymal stem cells with hialuronic acid according to the following scheme:

1. Group A: intra-articular injection of hyaluronic acid (Hyalone®). Single dose.
2. Group B: Low Dosage of MSCs . Intra-articular injection of 10 million autologous mesenchymal progenitor stem cells cultured ex - vivo (cell suspension sterile small volume (5-10 ml ) in a vehicle suitable for intraarticular injection ) followed by an intraarticular injection Hiaurónico Acid ( Hyalone®).
3. Group C : High dose of MSCs. Intra-articular injection of 100 million autologous mesenchymal progenitor stem cells cultured ex - vivo ( cell suspension sterile small volume (5-10 ml ) in a vehicle suitable for intraarticular injection ) followed by an intraarticular injection Hiaurónico Acid (Hyalone®).

The primary endpoint is safety and feasibility. The investigators registered the occurrence of complications and / or adverse effects during the study.

In addition the investigators assess the response to intra-articular infusion of CMM analyzing the following parameters:

* Clinical assessment of pain and function (Baseline, 1, 3, 6 and 12 months since treatment): VAS , WOMAC , KOOS , EuroQol, SF-16, Lequesne , WOMAC , KOOS.
* Radiographic (baseline, 6 and 12 months since treatment): Femorotibial space.
* Radiographic using MRI (baseline, 6 and 12 months since treatment): by assessing the number location of the lesions , cartilage thickness , signal intensity , subchondral bone alteration , volume and WORMS and dGEMRIC protocols.

DETAILED DESCRIPTION:
Purpose: To determine the safety, feasibility and effectiveness (clinical and radiological) of intra-articular administration of autologous mesenchymal stem cells (MSCs) in patients with knee osteoarthritis.

Patients and methods

Clinical trial phase I- II, randomized , multicenter , with three treatment arms and 10 patients for each group. The investigators compare the intraarticular injection of hialuronic acid against the administration of two different doses of mesenchymal stem cells with hialuronic acid according to the following scheme:

1. Group A: intra-articular injection of hyaluronic acid (Hyalone®). Single dose.
2. Group B: Low Dosage of MSCs . Intra-articular injection of 10 million autologous mesenchymal progenitor stem cells cultured ex - vivo (cell suspension sterile small volume (5-10 ml ) in a vehicle suitable for intraarticular injection ) followed by an intraarticular injection Hiaurónico Acid ( Hyalone®).
3. Group C : High dose of MSCs. Intra-articular injection of 100 million autologous mesenchymal progenitor stem cells cultured ex - vivo ( cell suspension sterile small volume (5-10 ml ) in a vehicle suitable for intraarticular injection ) followed by an intraarticular injection Hiaurónico Acid (Hyalone®).

The autologous mesenchymal stem cells are obtained from the iliac crest and cultured ex vivo under local anesthesia and sedation.

The primary endpoint is safety and feasibility. The investigators registered the occurrence of complications and / or adverse effects during the study.

In addition the investigators assess the response to intra-articular infusion of CMM analyzing the following parameters:

* Clinical assessment of pain and function (Baseline, 1, 3, 6 and 12 months since treatment): VAS , WOMAC , KOOS , EuroQol, SF-16, Lequesne , WOMAC , KOOS.
* Radiographic (baseline, 6 and 12 months since treatment): Femorotibial space.
* Radiographic using MRI (baseline, 6 and 12 months since treatment): by assessing the number location of the lesions , cartilage thickness , signal intensity , subchondral bone alteration , volume and WORMS and dGEMRIC protocols.

All patients met the following inclusion and exclusion criteria:

Inclusion Criteria:

* Males and females between 50 and 80 year old.
* Diagnosis of knee OA according to the criteria of osteoarthritis of the ACR (American College of Rheumatology).
* Joint pain equal or greater than 2.5 points on the visual analogue scale (VAS).
* Radiological Classification: Kellgren-Lawrence scale greater or equal to 2.
* Body mass index between 20 and 35 kg/m2.
* Ability to follow during the study period.

Exclusion Criteria:

* Bilateral Osteoarthritis of the Knee requiring treatment in both knees.
* Previous diagnosis of polyarticular disease.
* Severe mechanical deformation.
* Arthroscopy during the previous 6 months.
* Intraarticular infiltration of hyaluronic acid in the last 6 months.
* Systemic autoimmune rheumatic disease.
* Poorly controlled diabetes mellitus.
* Blood dyscrasias.
* Immunosuppressive or anticoagulant treatments.
* Treatment with corticosteroids in the 3 months prior to inclusion in the study.
* NSAID therapy within 15 days prior to inclusion in the study.
* Patients with a history of allergy to penicillin or streptomycin.
* Allergy to hyaluronic acid or poultry proteins.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 50 and 80 year old.
* Diagnosis of knee OA according to the criteria of osteoarthritis of the ACR (American College of Rheumatology).
* Joint pain equal or greater than 2.5 points on the visual analogue scale (VAS).
* Radiological Classification: Kellgren-Lawrence scale greater or equal to 2.
* Body mass index between 20 and 35 kg/m2.
* Ability to follow during the study period.

Exclusion Criteria:

* Bilateral Osteoarthritis of the Knee requiring treatment in both knees.
* Previous diagnosis of polyarticular disease.
* Severe mechanical deformation.
* Arthroscopy during the previous 6 months.
* Intraarticular infiltration of hyaluronic acid in the last 6 months.
* Systemic autoimmune rheumatic disease.
* Poorly controlled diabetes mellitus.
* Blood dyscrasias.
* Immunosuppressive or anticoagulant treatments.
* Treatment with corticosteroids in the 3 months prior to inclusion in the study.
* NSAID therapy within 15 days prior to inclusion in the study.
* Patients with a history of allergy to penicillin or streptomycin.
* Allergy to hyaluronic acid or poultry proteins.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Baseline Visual analogue scale (VAS) | prior to the initial dose on day 1
  Baseline Visual analogue scale (VAS)
Baseline value of knee injury and osteoarthritis outcome score (Koos). | Prior to the intervention on day 1
  Prior to the intervention on day 1 value of knee injury and osteoarthritis outcome score (Koos).
Baseline Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC). | Prior to the intervention on day 1
  Prior to the intervention on day 1 Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC).
Baseline SF-36 value | Prior to the intervention on day 1
  Prior to the intervention on day 1 SF-36 value
Baseline euroquol 5D value | Prior to the intervention on day 1
  Pretreatment euroquol 5D value
Baseline Lequesne index | Prior to the intervention on day 1
  Prior to the intervention on day 1 Lequesne index
Baseline femorotibial distance | Prior to the intervention
  Prior to the intervention femoritibial distance on rosenberg x-ray view
Number of Participants with Serious and Non-Serious Adverse Events Number of Participants with Serious and Non-Serious Adverse Events Number of Participants with Serious and Non-Serious Adverse Events | Follow up
  During the follow up
Visual analogue scale (VAS) at on month | 1 month
  Visual analogue scale (VAS) at on month
Visual analogue scale (VAS) at 3 months | 3 months
  Visual analogue scale (VAS) at 3 months
Visual analogue scale (VAS) at 6 months | 6 months
  Visual analogue scale (VAS) at 6 months
Visual analogue scale (VAS) at 12 months | 12 months
  Visual analogue scale (VAS) at 12 months
Value of knee injury and osteoarthritis outcome score (Koos) at 1 month | 1 month
  Value of knee injury and osteoarthritis outcome score (Koos) at 1 month
Value of knee injury and osteoarthritis outcome score (Koos) at 3 month | 3 Months
  Value of knee injury and osteoarthritis outcome score (Koos) at 3 month
Value of knee injury and osteoarthritis outcome score (Koos) at 6 month | 6 months
  Value of knee injury and osteoarthritis outcome score (Koos) at 6 month
Value of knee injury and osteoarthritis outcome score (Koos) at 12 months | 12 months
  Value of knee injury and osteoarthritis outcome score (Koos) at 12 months
Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC) at 1 month | 1 month
  Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC) at 1 month
Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC) at 3 month | 3 months
  Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC) at 1 month
Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC) at 6 month | 6 months
  Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC) at 6 month
Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC) at 12 months | 12 months
  Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC) at 12 months
SF-36 value at 1 month | 1 month
  SF-36 value
SF 36 value at 3 months | 3 months
  SF 36 value at 3 months
SF 36 value at 6 months | 6 months
  SF 36 value at 6 months
SF 36 value at 12 months | 12 months
  SF 36 value at 12 months
Euroquol 5D value at 1 month | 1 MOnth
  Euroquol 5D value at 1 month
Euroquol 5D value at 3 months | 3 months
  Euroquol 5D value at 3 months
Euroquol 5D value at 6 months | 6 months
  Euroquol 5D value at 6 months
Euroquol 5D value at 12 months | 12 months
  Euroquol 5D value at 12 months
Lequesne index at 1 month | 1 month
  Lequesne index at 1 month
Lequesne index at 3 months | 3 months
  Lequesne index at 3 months
Lequesne index at 6 months | 6 months
  Lequesne index at 6 months
Lequesne index at 12 months | 12 months
  Lequesne index at 12 months
Femorotibial distance at 6 months | 6 months
  Femorotibial distance at 6 months
Femorotibial distance at 12 months | 12 months
  Femorotibial distance at 12 months
Baseline MRI WORMS protocol | Prior to the intervention
  Prior to the intervention MRI WORMS protocol
MRI WORMS protocol score at 6 months | 6 months
  MRI WORMS protocol score at 6 months
MRI WORMS protocol score at 12 months | 12 months
  MRI WORMS protocol score at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: José Lamo-Espinosa, MD, Principal Investigator — Clinica Universidad de Navarra; Felipe Prosper, MD PhD, Study Director — Clinica Universidad de Navarra; Juan Blanco, MD PhD, Principal Investigator — University of Salamanca
Locations (2):
- Spain (2):
  - Traumatology department. Complejo Hospitalario de Salamanca, Salamanca, Castille and León
  - Orthopaedic and traumatology department. Clínica Universidad de Navarra, Pamplona, Navarre

REFERENCES:
- [Derived] Lamo-Espinosa JM, Prosper F, Blanco JF, Sanchez-Guijo F, Alberca M, Garcia V, Gonzalez-Vallinas M, Garcia-Sancho J. Long-term efficacy of autologous bone marrow mesenchymal stromal cells for treatment of knee osteoarthritis. J Transl Med. 2021 Dec 11;19(1):506. doi: 10.1186/s12967-021-03160-2. PMID 34895259
- [Derived] Lamo-Espinosa JM, Mora G, Blanco JF, Granero-Molto F, Nunez-Cordoba JM, Lopez-Elio S, Andreu E, Sanchez-Guijo F, Aquerreta JD, Bondia JM, Valenti-Azcarate A, Del Consuelo Del Canizo M, Villaron EM, Valenti-Nin JR, Prosper F. Intra-articular injection of two different doses of autologous bone marrow mesenchymal stem cells versus hyaluronic acid in the treatment of knee osteoarthritis: long-term follow up of a multicenter randomized controlled clinical trial (phase I/II). J Transl Med. 2018 Jul 31;16(1):213. doi: 10.1186/s12967-018-1591-7. PMID 30064455
- [Derived] Lamo-Espinosa JM, Mora G, Blanco JF, Granero-Molto F, Nunez-Cordoba JM, Sanchez-Echenique C, Bondia JM, Aquerreta JD, Andreu EJ, Ornilla E, Villaron EM, Valenti-Azcarate A, Sanchez-Guijo F, Del Canizo MC, Valenti-Nin JR, Prosper F. Intra-articular injection of two different doses of autologous bone marrow mesenchymal stem cells versus hyaluronic acid in the treatment of knee osteoarthritis: multicenter randomized controlled clinical trial (phase I/II). J Transl Med. 2016 Aug 26;14(1):246. doi: 10.1186/s12967-016-0998-2. PMID 27565858
- See also: University clinic of navarre trial information — http://www.cun.es/actualidad/noticias/celulas-madre-osea-artrosis-rodilla